# Research protocol 4th National Registry of Cardiovascular Surgery (CCV) in Argentina

*-Version N ° 3- 8 of JULY 2021* 


2

Confidentiality notice: The concepts and information included in this document are confidential and exclusive and not

they must be disclosed in whole or in part without the express written consent of the coordinator.


3

## PROTOCOL SUMMARY

#### ➤ Title

1- Prospective registry of patients undergoing CCV in Argentina

#### ➤ Study Phase

1- Prospective Registry (IV)

#### ➤ Evaluation

1- Follow-up of patients during hospitalization and 30 days after surgery.

#### > Primary Objectives

1.a.

Determine the evolution and surgical complications in patients undergoing CCV

To determine the association between different risk variables during the intranosocomial stay and at 30 days of discharge including nosocomial readmission during the 30-day follow-up.

#### > Secondary Objectives

To determine the association between different variables that occurred before, during and after the surgical intervention.

To determine the association between different variables of risk at discharge and the rate of complications, including

mortality and readmissions during the 30 days following discharge, such as:

Cardiovascular mortality, all-cause mortality, rehospitalization, infectious complications.

To determine the association between different variables with cardiovascular mortality in relation to CCV.

Assess eventual complications 30 days after hospital discharge


4

#### ➤ Study Design

National, multicenter, analytical, prospective cohort study for prognostic evaluation in patients undergoing

cardiovascular surgery (CCV)

#### ➤ Sample Size

The largest number of patients (between 2000 and 3000) will be enrolled during a set period of time (1 year), from

October 1, 2020 to September 30, 2021

#### ➤ Eligibility Criteria

Over 18 years

Г

| Myocardial revascularization surgery |
|---|
| Valvular surgeries |
| A coording A ortio Surgary |
| Ascending Aortic Surgery |
| Type A Aortic Dissection Surgery |
| Type A Aorne Dissection Surgery |
| Combined surgery |
| ➤ Exclusion Criteria |
| Cardiovascular surgery for congenital pathologies |
| Peripheral vascular surgery |
| Cardiovascular surgery secondary to trauma |
| Thoracic and abdominal aorta pathology |
| Other surgeries |
| ➤ Procedures |
| Various centers are included nationwide with a CCV service capable of admitting and intervening |
| patients with |
| criteria already established. |
| They are arranged below: |
| Leben Health |
| Private Hospital Santa Clara de Asis |
| Dr Alberto Duhau Hospital Pasteur Clinic |
| Sanatorio Juan XXIII |
| Private hospital |
| San Martin Sanatorium |
| Cordoba Hospital |
| Spanish Hospital |
| Spanish Hospital / Pami 2 Polyclinic / Italian Hospital / IPAM |
| Santa Clara Clinic |
| CARDIOMED |
| Cosme Argerich Hospital |
| Spanish Society of Mutual Aids |
| CCV- St. Clara San Juan |
| P |


5

Tucuman Institute of Heart Diseases

Italian Hospital of Mendoza

FIG Dr. Oscar Alende

HOSPITAL FOUNDATION / CENTRAL MILITARY HOSPITAL

Spanish Hospital

Galen Sanatorium

San Juan de Dios Hospital

Guemes sanatorium

Dr. Cesar Milstein Hospital

CEMIC

HIEAYC SAN JUAN DE DIOS

Sanatorio de la Cañada

Hospital de Clinicas Jose de San Martin

South Mendocino Spanish Hospital

Sanatorium of La Trinidad Miter

La Sagrada Familia Clinic

**ICBA** 

Santorio de la Trinidad Quilmes

British Sanatorium of Rosario

Bazterrica

Santa Isabel Clinic

Htal Churruca

Sanatorio Del Salvador

Sanatorio Anchorena San Martin

Carrillo Hospital

Sanatorium San Juan Bautista

Sanatorio Juan XXIII

Sanatorio Juan XXIII

Argerich Hospital

Argerich hospital

HIGA President Peron

Spanish Hospital Buenos Aires

Belgrano Adventist Clinic

German Hospital

Syrian Lebanese Hospital

BRITISH Hospital

Favaloro Foundation

Private Clinic velez sarsfield

Yunes Clinic

Hospital Italiano De Bs.As.

Juan Domingo Peron High Complexity Hospital

Allende Sanatorium

Sanatorio de la Cañada

Cardiology institute

British sanatorium

Htal Eduardo Wilde

Presidente Peron Hospital

Hospital El Cruce

Private hospital

Pasteur Clinic

Hospital Escuela de Agudos Ramon Madariaga

Bernal Sanatorium

San Roque Sanatorium

Spanish society and clinic santa clara mendoza


6

Cesar Milstein Hospital

San Luis Cardiovascular Institute

Galen Sanatorium

**ICBA** 

Instituto de Cardiologia de Rosario "Dr. Luis Gonzalez Sabathie"

Malvinas Argentinas Sanitary Pole

Delta Sanatorium

Sanatorio Dr Julio Mendez

Model Institute of Cardiology

Sanatorio San Jorge SRL

policlinico san lucas / clinica regional del sud

Private Hospital of the Mar del Plata Community

SANTA FE SANATORIO MEDICO SURGICO

Zabala SMG Clinic

Decentralized Public Hospital Dr Guillermo Rawson

Patients are evaluated during hospitalization eligibility criteria and the Informed Consent will be signed. (CI) according to current regulations.

The respective filling of the files designed with the necessary Pre-surgical data will be carried out, during the

surgical procedure and postoperative.

Telephone calls will be made from the Argentine Society of Cardiology (SAC) and / or College of Cardiovascular Surgeons (CCV), with a questionnaire 30 days after discharge.

The principal investigators of the study are:

Dr Esteban Romeo

Dr Adrián Lescano

It will be assigned during the inclusion of investigator patients for each of the centers, who will be responsible for completing the form ( *CRF* ) and sending the registered data.


7

# Additional Information

#### Introduction

More than ten years have passed since the last CCV registration in the Argentine Republic In recent decades, the evolution of CCV has shown a reduction in the rate of complications and mortality in centers specialized

#### objectives

#### Record

- 1. determine complications, mortality and hospital stay, as well as evolution at 30 days after CVD In our country
- 2. Compare our variables with those exposed by the different international scores and thus be able to predict the

estimated evolution of our patients.

#### Substudy

1. Determine the association between different variables, complication rate and mortality 30 days after discharge.

# Proposed design

The study consists of **2 stages**, with the voluntary participation of the different centers, which is divided into nosocomial phase and phase a

30 days after discharge

Prospective multicenter registry of prognostic correlation with various risk scores in patients undergoing CCV and

evolution of the same 30 days after discharge

### Material and methods

Patients who meet the eligibility criteria described above are included from October 1, 2020 The protocol consists of 2 stages:

1) Nosocomial Phase: a descriptive record is made of the referred variables and the risk parameters upon discharge from

the patients

2) 30 days after discharge, the respective forms will be filled out for the final evaluation of patients who have undergone CCV and discharged from participating institutions


8

# Specific Protocol (Operational Definition of Variables):

A complete clinical history of the patient is taken (according to usual practice) and the data is filled out in the Pre, Intra and Post-surgical stage according to what is established in the form

# Affiliate Information and Background

Syncope Yes No SAHOS Yes No COPD No Mild Moderate Severe It is unknown

| Record ID | and background |
|---|---|
| Date of admission | |
| Acronyms for Name and Surname | |
| Last 3 digits of document number (Last 3 digits only) AgegenderWeight (kg) Public Hospital Coverage PAMI Social work Prepaid Particular Telephone Phone 2 Email Background Arterial hypertension Yes No Diabetes Yes No Diabetic retinopathy Yes No Dyslipidemia Yes No Ex-smoker tobacco I never smoke Smokes daily Smokes occasionally It is unknown | |
| | Height (cm) |
| 9 Hyperuricemia Yes No HIV Yes No Systolic LV dysfunction Yes No Heart failure Yes No Myocardial infarction No <30 days> 30 day Myocardial revascularization surgery Yes No Valve surgery Yes No Other cardiovascular surgery Yes No Type of cardiovascular surgery (Describe) Coronary angioplasty Yes No Immunocompromise Yes No Mediastinal radiation Yes No Stable chronic angina Yes No Chronic atrial fibrillation Yes No Unstable angina Yes No Family history of coronary disease Yes No Peripheral vascular disease Yes No Pulmonary Hypertension Yes No Cerebrovascular disease Yes No | |

Remote Non-Recent Pneumonia

It is unknown

Did you have COVID-19 within the month prior to surgery? If not

Liver disease Yes No

Illicit drug use No Recent Remote

It is unknown

Alcohol abuse No

<1 glass per day

2 to 7 glasses per day

> 7 glasses per day

It is unknown

Usual medication Aspirin


10

Clopidogrel

Ticagrelor

Prasugrel

Statins

Beta-blockers

**ACEI** 

ARA-II

Loop diuretics

Thiazides

Spirinolactone

Insulin

Oral hypoglycemic

Anticoagulants

Suspension P2Y12 Inhibitors Yes No

Days of suspension of Inhibitors P2Y12

Frail patient Yes No

I use a fragility score Yes No

Fragility score

Other background

Presurgical data

Presurgical diagnosis Heart failure

Endocarditis

Acute aortic syndrome

Ischemic heart disease

Valvular disease

Pericardial involvement

Other

Related signs and symptoms Dyspnoea

Precordial pain

Edema in lower limbs

Febrile syndrome

Syncope

Palpitations

Neurological focus

Acute Pulmonary Edema

Tachyarrhythmias

Bradyarrhythmias

Other


eleven

(Select at least one)

Coronary heart disease Yes

No

Left Coronary Trunk Injury Yes

| M. |
|---|
| No<br>Number of glasses |
| Vessels affected Descending Anterior |
| Diagonal Circumflex |
| Lateroventricular |
| Right Coronary |
| Other |
| Valvular disease Yes |
| No |
| Type of valve pathology Aortic stenosis |
| Aortic insufficiency Mitral stenosis |
| Mitral Insufficiency |
| Pulmonary stenosis |
| Pulmonary insufficiency |
| Tricuspid stenosis |
| Tricuspid Insufficiency |
| (Select at least one) |
| Combined Surgery Yes |
| No<br>(Valular + Bridges) |
| Type of procedure Scheduled |
| Urgency |
| Emergency |
| Laboratory upon admission |
| Hematocrit Leukocytes Platelets |
| Blood glucose Uremia Creatinine |
| Cholesterol HDL LDL Triglycerides Total bile GOT |
| GPT |
| Electrocardiogram |
| Rhythm Frequency |
| Prolonged PR AV block |
| Right bundle branch block Left bundle branch block |
| ST elevation ST elevation |
| 12 |
| T wave inversion |
| SCORES |
| We ask you to complete the following values by calculating them. Click on the following links to |
| enter the respective online calculators: |
| EUROSCORE: https://www.rccc.eu/Cardio/euroscoreII.html |
| ARGENSCORE: http://argenscore.org/calculadora.aspx EUROSCORE II mortality (%) |
| ARGENSCORE score |
| ARGENSCORE Mortality |
| Use of pre-surgical IACB Yes No |
| Use of Swan Ganz presurgical Yes No |
| Use of presurgical inotropics Yes No |
| Intraoperative |
| Date of surgery |
| Patient condition Stable Unstable |
| Use of ventricular assist Yes No |
| Use of BCIAo Yes No |
| Required transfusion of blood products Yes No |
| Red blood cells |
| (Units) |
| Platelets |
| (Units) |

#### Plasma

(Units)

Extracorporeal circulation Yes No

CEC time

(Minutes)

Clamping time

(Minutes)

CRM was carried out Yes No

Left breast bridge Yes No

Right breast bridge Yes No

Radial bridge Yes No

Number of radial bridges


13

Venous bridge Yes No

Number of venous bridges

Endarterectomy Yes No

Quality of the distal beds Good Regular

Bad

Valve surgery was performed Yes No

Aortic valve plastic Yes No

Aortica Jacoub plastic technique

David

Aortic valve replacement Yes No

Type of Biological Aortic Valve with stent

Biological without stent

Single Disc Mechanics

Clamshell Mechanics

Biological valve type Aortic Pericardial

Swine

Bovine

Aortic biological valve measurement

(Number)

Brand of Aortic Biological Valve

Aortic mechanical valve measurement

(Number)

Aortica mechanical valve brand

Ring enlargement Yes No

Ring enlargement technique

Plastic Mitral Valve Yes No

Plastic was made on the previous valve

Posterior leaflet

Mitral valve replacement Yes No

Biological Mitral Valve Type with Stent

Biological without stent

Single Disc Mechanics

Clamshell Mechanics

Type of Mitral Pericardial Biological Valve

Swine

Mitral biological valve measurement

(Number)

Mitral Biological Valve Brand

Mitral mechanical valve measurement

(Number)

Mitral mechanical valve brand

Intra-operative TEE in mitral surgery Yes No Plastic Tricuspid Valve Yes No Tricuspid valve replacement Yes No Biological Tricuspid Valve Type Mechanics

Tricuspid biological valve measurement

(Number)

Brand of Tricuspide Biological Valve

Tricuspid mechanical valve measurement

(Number)

Tricuspid mechanical valve brand

Pulmonary valve plastic Yes No Pulmonary valve replacement Yes No Biological Pulmonary Valve Type Mechanics

Pulmonary biological valve measurement

(Number)

Pulmonary biological valve brand

Pulmonary mechanical valve measurement

(Number)

Pulmonary mechanical valve brand

Ross Surgery Yes No


#### fifteen

Ascending Aortic Surgery Yes No Type of Ascending Aorta Surgery Bentall de Bono

Daguenancian

Resuspension

WHEAT (supracoronary)

Tirone David

Yacoub

Cabrol

Tubular portion replacement

Reattachment of supra-aortic vessels

Other

Aortic prosthesis placement Yes No

Aortic prosthesis measurement

(Number)

Intra-surgical hemorrhage Yes No Cause of Medical Surgical Bleeding Intra-surgical arrest Yes No Readmission to CEC Yes No

Other complications

# Postoperative

Via air Fast track (extubate)

Intubated Extubates at <6 hours 6 to 12 hours 12 to 24 hours > 24 hours Long ARM Yes No ARM days

Reintubation Yes No

Hemorrhage Yes No

(> 500 ml in the 1st hour or> 400 ml in the 2nd hour or

> 300 ml in the 3rd hour or> 200 ml in the 4th hour or

> 100 ml in the 5th hour)

Type of Hemorrhage Medical Surgical

Surgical examination required Yes No

Surgical resolution Yes No

Transfusion of blood products Yes No

Right Ventricular Dysfunction Yes No

(Persistent arterial hypotension, blood pressures

#### Page 16

#### 16

Elevated ventricular (right atrium) filling,

low cost with need for intervention

pharmacological and eventually mechanical (TAPSE <17

mm or visual impression by Echocardiography of

RV dysfunction))

Low expenditure syndrome Yes No

(Systolic blood pressure <90 mmHg, pale and

skin coldness, lack of capillary filling,

clouding and oliguria, heart index

< 2.2

L / min / m2, pulmonary capillary pressure> 18 mmHg, with

inotropic and / or balloon requirement

intra-aortic counterpulsation (IACAB))

Inotropic / vasopressor requirement Yes No

Inotropics / Vasopressors used Dopamine

Dobutamine

Milrinone

Levosinmendan

Noradrenaline

Vasopressin

Adrenalin

Swan Ganz requirement Yes No

Perioperative myocardial infarction Yes No

Definition of perioperative infarction according to the center Development of Q waves

per ... Increased CPK MB â ‰ ¥ 80 IU / ml

Parietal alterations on echocardiogram

Troponin T or I> 10 times its baseline value

US troponin> 10 times baseline

Atrial fibrillation Yes No

Atrioventricular block Yes No

Complex ventricular arrhythmia Yes No

Transient pacemaker Yes No

Permanent pacemaker Yes No

I do prophylaxis for postoperative AF Yes No

Drug used

POP day of initiation of prophylaxis for AF

Renal failure Yes No

(Increase in creatinine above 50%

with respect to the baseline value and / or

17

hemodialysis)

Hemodialysis Yes No

Stroke Yes No

(Focal and / or diffuse brain injury confirmed by

clinical findings and / or computed tomography with

sensory or motor sequelae upon discharge of the patient)

Transient ischemic accident Yes No

Psychiatric disorders Yes No

(Any of the following: delirium, hallucinations,

psychomotor arousal)

Required treatment with ... Risperidone

Quetiapine

Haloperidol

Other

Respiratory distress syndrome Yes No

(Infiltrate in 4 quadrants - PCP <18 - PAFI <200)

Fever without obvious focus Yes No

Sepsis Yes No

(Suspected or documented infection with dysfunction of

target organ and at least two of the following

criteria: Temperature> 38 Â ° C or <36 Â ° C,

White blood cell count greater than 12,000 uL or less

at 4000 uL, Tachycardia, Tachypnea> 30 rpm,

Altered mental state, Positive culture of

primary focus of infection, mean arterial pressure

less than 70 mm Hg for a minimum

fingers

hours, poor distal perfusionâ € ")

Urinary infection Yes No

Respiratory infection Yes No

Surgical wound infection Yes No

Superficial wound infection Yes No

Saphenous wound infection Yes No

Sternal infection Yes No

Mediastinitis Yes No

Sternal reopening requirement Yes No

Sternal reopening POP day

Sternal mechanical instability Yes No

COVID-19 infection development during internment


18

If not

TOTAL days of hospitalization until discharge

POSTOPERATIVE days until discharge

Discharge

Alive

Dead

Death cause:

Infectious

Cardiovascular

Distributive shock

Hemorrhage

Cardiac tamponade

Stroke

Respiratory distress

Multi-organ failure

Another cause

Death from infectious cause: Mediastinitis Pneumopathy Sepsis Other

| Identified germ |
|---|
| Death from cardiovascular cause: Myocardial infarction Arrhythmia Heart failur |
| Pre Registration Laboratory |
| Hematocrit Blood glucose |
| Uremia Creatinine |
| Medication at discharge ASA |
| Clopidogrel |
| Ticagrelor |
| Prasugrel |
| Statins |
| Beta-blockers |
| Sartan |
| ACE inhibitors |
| Loop diuretic |
| Thiazide |
| Spironolactone |
| Insulin |
| Oral hypoglycemic |
| Anticoagulants |
| Investigator Notes |


19

# Follow-up

Re-internment Yes No

(Within the first 30 days after discharge)

Cause of re-admission:

Heart failure

Respiratory insufficiency

Renal insufficiency

Sepsis:

Other

Sepsis Yes: Sepsis starting point: Mediastinitis or other focus

Another cause of re-admission

Death no

Death Yes:

(Within the first 30 days after discharge)

Cause of death in follow-up: Cardiovascular- NON-cardiovascular cause

\_\_\_\_\_